CLINICAL TRIAL: NCT06249009
Title: Impact of Increasing Flow Rates in High-flow Nasal Cannula and CPAP on Diaphragmatic Work in Newborn and Paediatric Population: Non-inferiority Study
Brief Title: Diaphragmatic Work During HFNC and CPAP Support
Acronym: DiaWorkHFNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Maquet Critical Care AB (Industry); Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AOI 2022 SAVY
Record Dates: First submitted 2023-09-28; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-06

CONDITIONS: Respiratory Insufficiency in Children; Newborn Rds; Nasal Cannula; CPAP Ventilation
Keywords: Paediatric; HFNC; CPAP; work of breathing; primary support
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The included patients will then be randomized into two separate groups: a CPAP group with PEEP at 7 cmH2O for 30 minutes and an HFNC group with increasing flow rates from 2L/kg/min to 5 L/kg/min with 30 minutes of study for each flow. After a wash-out period of 15 minutes, according to the cross-over procedure, the patients will change groups in order to perform the remaining analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP-first group (Active Comparator): After a wash out of 15 minutes with conventional oxygen therapy, CPAP with a Positive End -Expiratory Pressure of 7 cmH2O will be introduced, with an inspiratory oxygen fraction required for an oxygen saturation of 94%, during 30 minutes. The collection of EAdi min/max will be done every minutes over 30min as well as the collection of HR, Respiratory rate (RR), SpO2, while TCPCO2, distress respiratory score and pain score will be taken at M0 and M30.
  Interventions: Device: Non invasive ventilation
- HFNC-first group (Active Comparator): After a wash out of 15 minutes with conventional oxygenotherapy, increasing flow rates for up to 2 hours according to the following augmentation:
  * Initiation at a flow rate of 2 L/kg/min with FiO2 required to achieve SpO2≥94% (increase FiO2 if reliable SpO2 signal <94% for 1 minute) for 30min.
  * Increase to 3 L/kg/min after the first 30min of ventilation and repeat the previously described experimental scheme.
  * Further increase to 4 L/kg/min after 30min of ventilation and repetition of the experimental scheme (if weight < 16 kg).
  * Last increase to 5 L/kg/min after 30 min of ventilation and repetition of the experimental scheme (if weight < 13 kg).
  The collection of EAdi min/max will be done every minutes over 30min as well as the collection of HR, RR, SpO2, while TCPCO2, distress respiratory score and pain score will be taken at M0 and M30.
  Interventions: Device: Non invasive ventilation

INTERVENTIONS:
Device: Non invasive ventilation — CPAP and increasing flows of HFNC will be compared during a 30-minutes period each

SUMMARY:
The goal of this randomised controlled, cross-over clinical trial is to compare High Flow Nasal Cannulas (HFNC) and Continuous Positive Airways Pressure (CPAP) in neonates over 34 weeks' amenorrhoea (SA) up to children weighing less than 20 kg with respiratory failure.

The main question it aims to answer is the non-inferiority of high flows of high-flow nasal cannula compared with CPAP by analysis of diaphragmatic contraction (EAdi (Electrical activity of diaphragm)).

Participants with respiratory failure and need of non invasive ventilation and nasogastric tube will receive 4 different increasing flows of HFNC and Positive End-Expiratory Pressure of 7 cmH2O with CPAP during 30 minutes for each flow rate and CPAP. The electrical activity of diaphragm and clinical data of the patient upon each flow and support will be collected. According to the cross-over procedure, the patients will change groups (increasing flows of HFNC or CPAP) in order to perform the remaining analysis.

DETAILED DESCRIPTION:
With this research protocol, the investigators aim to demonstrate the non-inferiority of high flows of HFNC compared with CPAP on work of breathing (based on the intensity of contraction of diaphragmatic fibres and clinical aspects) in paediatric and neonatal patients. The investigators will also study the clinical tolerance and safety of these practices.

Objectives :

Main objective: To demonstrate the non-inferiority of high-flow nasal cannula flow rates compared with CPAP by analysis of diaphragmatic contraction (EAdi (Electrical activity of diaphragm)) in neonates over 34 weeks' amenorrhoea (SA) up to children weighing less than 20 kg in respiratory failure.

Secondary objectives:

* To compare different flows of HFNC (2 L/kg/min, 3 L/kg/min, 4 L/kg/min, 5 L/kg/min) with each other by analysing diaphragmatic contraction.
* Compare the clinical effectiveness of different flow rates of HFNC with CPAP in young children in respiratory distress.
* To compare the tolerability of different flow rates of HFNC with CPAP in the population of young children suffering from respiratory distress.
* To compare the incidence of minor (digestive discomfort, digestive bloating, non-damaging skin lesions) and major (thoracic barotrauma, damaging skin lesions) side effects of different flow rates of HFNC with CPAP in young children in respiratory distress.
* To describe the choice of support and settings (flow rates or PEEP levels) made by the practitioners in charge of the child after the study period.
* To describe the epidemiological data from the paediatric intensive care and monitoring units and the neonatal intensive care unit.

Type of study: Randomised controlled, cross-over, single-centre, non-inferiority trial of a medical device.

Number of centres: 1

Study design:

Upon admission to the department, if the eligibility criteria are met and the parents agree to the research , a wash-out period will be performed under low-flow oxygen therapy at 1 L/min to achieve SpO2 ≥ 94% for 15 minutes.

The included patients will then be randomized into two separate groups: a CPAP group with PEEP at 7 cmH2O for 30 minutes and an HFNC group with increasing flow rates for up to 2 hours.

The patients included will be their own controls and at the end of the first analysis, according to the cross-over procedure, the patients will change groups in order to perform the remaining analysis.

A recourse procedure has been foreseen in case of failure of ventilatory support.

Medical devices :

Concerning HFNC ventilation:

The nasal cannulas used are Optiflow® cannulas (Fisher and Paykel Laboratory) which will be adapted to the size of each patient's nostrils. The following sizes are available:

* NICU patient: Optiflow Junior 2®.
* PICU patient: Optiflow Junior 2®, Optiflow +®.

Concerning CPAP ventilation:

* For the neonatal population:

  * Medin Sindi® CPAP masks, caps and ties
  * Medin Miniflow® CPAP generators
* For the paediatric population :

  * Medin Sindi® CPAP masks, caps and ties
  * Fisher and Paykel Healthcare CPAP masks, cannulas and caps
  * Miniflow® CPAP generators from Medin
  * Fisher and Paykel Healthcare CPAP generators

Expected benefits :

If it is shown that a reduction in the work of breathing is observed (EAdi and usual clinical signs) when HFNC flow rates are gradually increased, and that this increase to flow rates of 3 to 5 L/kg/min is well tolerated and does not increase the risk of barotrauma, HFNC ventilation at flow rates greater than 2 L/kg/min could be more widely proposed and accepted in the various units using it, as it is unanimously accepted in terms of tolerance and comfort for the patient compared with CPAP.

Recruitment procedures The patients eligible for this study will be those admitted to the neonatal and paediatric intensive care unit of the Clermont-Ferrand University Hospital by a doctor on the unit and who meet the various inclusion criteria for the study.

An information note has been drawn up and will be presented and explained to the child's legal representative(s) by an investigating doctor during their usual care, as well as to the child if his or her level of understanding is adequate, within 2 hours of admission to the department. The parents and the child will have a maximum of 1 hour to reflect (and a maximum of 3 hours from admission to the ward) between the time they are given the information and the time they sign the consent form.

Legal representative(s) will then be asked to sign the written consent. The child's inclusion in the DiaworkHFNC protocol will be recorded in the child's computerised medical record (ICCA software).

ELIGIBILITY:
Inclusion Criteria:

* Newborns over 34 SA and paediatric patients weighing less than 20 kg.
* Need for ventilatory support by HFNC or CPAP for respiratory failure
* Need for enteral feeding via nasogastric tube
* Hospitalized in PICU or NICU at Clermont-Ferrand University Hospital,
* Covered by Social Security.
* Whose parents or guardians are able to provide informed consent to participate in the research.

Exclusion Criteria:

* Respiratory failure requiring immediate intubation.
* Use of HFNC or CPAP as a relay to extubation.
* Acquired or congenital abnormality of the gastrointestinal tract.
* Diaphragmatic paralysis and/or neuromuscular pathology
* Failure of central ventilatory control (e.g. intra-ventricular haemorrhage, anoxic-ischaemic encephalopathy, massive vascular accident, intracranial process, cerebral edema and/or intracranial hypertension).
* Contraindications listed in the CPAP and HFNC user manuals: absence of spontaneous ventilation, choanal atresia, diaphragmatic hernia, tracheo-oesophageal fistula, nasal trauma, severe deformity likely to be aggravated by the nasal mask or nasal cannula, pneumothorax, pneumencephaly, Cerebrospinal Fluid leak, hypotension.
* Refusal by parents or guardians.

Ages: 34 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-11-27 (Estimated); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Variations of mean max electrical activity of the diaphragm (mean EAdi) between different HFNC flows and between each HFNC flow and CPAP | Maximal electrical activity of diaphragm will be recorded every minutes (up to 3 hours)
  Maximal EAdi will be measured in µV

SECONDARY OUTCOMES:
Variation in mean minimum EAdi (EAdi min) between different HFNC flows and between each HFNC flow and CPAP | Minimal electrical activity of diaphragm will be recorded every minutes (up to 3 hours)
  Minimum EAdi will be measured in µV
Variations of heart rate between the different rates of HFNC and between each rate of HFNC and CPAP | every 5 minutes during 3 hours
  Heart rate will be measured in beats per minute (bpm)
Variations of respiratory rate between the different rates of HFNC and between each rate of HFNC and CPAP | every 5 minutes during 3 hours
  Respiratory rate will be measured in breath per minute
Variations of oxygen saturation between the different rates of HFNC and between each rate of HFNC and CPAP | every 5 minutes during 3 hours
  Oxygen saturation will be measured in percentage
Variations of transcutaneous partial pressure of carbon dioxide between the different rates of HFNC and between each rate of HFNC and CPAP | every 5 minutes during 3 hours
  Transcutaneous partial pressure of carbon dioxide will be measured in mmHg
Variations of respiratory distress score between the different rates of HFNC and between each rate of HFNC and CPAP | Every 30 minutes during 3 hours
  score of Silverman (0 to 10), or score modified Wood score (0 to 10) or score of PRAM (0 to 12) depending on the pathology
Incidence of minor side effects for each HFNC flow rate and for CPAP | Every 30 minutes during 3 hours
  bloating and/or gastrointestinal discomfort with no other associated cause, low-grade skin trauma
Incidence of major side effects for each flow of HFNC and for CPAP | Every 30 minutes during 3 hours
  Barotrauma to the chest, pneumothorax or pneumomediastinum
  Bradycardia defined as :
  if < 1 year: Heart rate (HR) < 100 bpm for 20 seconds or < 60 bpm for 5 seconds if ≥ 1 year: HR < 100 bpm for 20 seconds or < 40 bpm for 5 seconds Number of desaturations (oxygen saturation rate (SpO2) < 88% for 3s), apneas (breathing pause ≥ 10s) High-grade skin trauma
Intubation rate | through patient follow-up period, up to 3 hours
Ventilatory weaning time | From date of randomization until the date of pressure weaning support, up to 30 days.
  Weaning from all types of pressure support

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Savy, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramnarayan P, Richards-Belle A, Drikite L, Saull M, Orzechowska I, Darnell R, Sadique Z, Lester J, Morris KP, Tume LN, Davis PJ, Peters MJ, Feltbower RG, Grieve R, Thomas K, Mouncey PR, Harrison DA, Rowan KM; FIRST-ABC Step-Up RCT Investigators and the Paediatric Critical Care Society Study Group. Effect of High-Flow Nasal Cannula Therapy vs Continuous Positive Airway Pressure Therapy on Liberation From Respiratory Support in Acutely Ill Children Admitted to Pediatric Critical Care Units: A Randomized Clinical Trial. JAMA. 2022 Jul 12;328(2):162-172. doi: 10.1001/jama.2022.9615. PMID 35707984
- [Result] Milesi C, Essouri S, Pouyau R, Liet JM, Afanetti M, Portefaix A, Baleine J, Durand S, Combes C, Douillard A, Cambonie G; Groupe Francophone de Reanimation et d'Urgences Pediatriques (GFRUP). High flow nasal cannula (HFNC) versus nasal continuous positive airway pressure (nCPAP) for the initial respiratory management of acute viral bronchiolitis in young infants: a multicenter randomized controlled trial (TRAMONTANE study). Intensive Care Med. 2017 Feb;43(2):209-216. doi: 10.1007/s00134-016-4617-8. Epub 2017 Jan 26. PMID 28124736
- [Result] Milesi C, Pierre AF, Deho A, Pouyau R, Liet JM, Guillot C, Guilbert AS, Rambaud J, Millet A, Afanetti M, Guichoux J, Genuini M, Mansir T, Bergounioux J, Michel F, Marcoux MO, Baleine J, Durand S, Durand P, Dauger S, Javouhey E, Leteurtre S, Brissaud O, Renolleau S, Portefaix A, Douillard A, Cambonie G; GFRUP Respiratory Study Group. A multicenter randomized controlled trial of a 3-L/kg/min versus 2-L/kg/min high-flow nasal cannula flow rate in young infants with severe viral bronchiolitis (TRAMONTANE 2). Intensive Care Med. 2018 Nov;44(11):1870-1878. doi: 10.1007/s00134-018-5343-1. Epub 2018 Oct 21. PMID 30343318
- [Result] Nasef N, El-Gouhary E, Schurr P, Reilly M, Beck J, Dunn M, Ng E. High-flow nasal cannulae are associated with increased diaphragm activation compared with nasal continuous positive airway pressure in preterm infants. Acta Paediatr. 2015 Aug;104(8):e337-43. doi: 10.1111/apa.12998. Epub 2015 Apr 13. PMID 25759095
- [Result] Pham TM, O'Malley L, Mayfield S, Martin S, Schibler A. The effect of high flow nasal cannula therapy on the work of breathing in infants with bronchiolitis. Pediatr Pulmonol. 2015 Jul;50(7):713-20. doi: 10.1002/ppul.23060. Epub 2014 May 21. PMID 24846750